CLINICAL TRIAL: NCT03435705
Title: Maintenance of Occupational Therapy for Patients With Alzheimer: A Pragmatic Randomized Trial
Brief Title: Maintenance of Occupational Therapy for Patients With Alzheimer
Acronym: MaTheoAlz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CHUBX 2016/29
Record Dates: First submitted 2018-01-18; First posted 2018-02-19 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Alzheimer's Disease or Related Disorder
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention arm (Experimental): maintaining of occupational therapy for a 4 months period
  Interventions: Behavioral: maintaining of occupational therapy
- control arm (No Intervention): usual care after the end of the recommended initial program

INTERVENTIONS:
Behavioral: maintaining of occupational therapy — 8 home sessions over a 4 months period with caregivers' education, occupational therapy and care coordination for post intervention
  Arms: intervention arm

SUMMARY:
France put a massive effort for improving dementia care through a national Alzheimer plan in 2008 and this effort was confirmed by the next government (Neurodegenerative Diseases Plan 2014-2019). Some new care models and interventions have been implemented such as Alzheimer specialized teams offering occupational therapy. The teams intervene at home with medical prescription. A recent pilot study demonstrated that occupational therapy has the potential to bring clinical benefits for both dementia patients and their caregivers. Nevertheless, occupational therapy has been designed as a short-term intervention and the end of intervention is challenging for therapists and patients. We aim to test the clinical and economic efficacy of maintaining occupational therapy over supplementary 4 months in a pragmatic randomized controlled trial.

DETAILED DESCRIPTION:
The Alzheimer specialized teams provide "occupational" therapy to maintain or restore the functional capacities of patients. After a deep evaluation of the expectations and needs of patients and their caregivers, the therapists propose to work one or more specific activities that were once pleasant through 12 to 15 sessions at home over 3 months. They also advise individuals to optimize home safety. A pilot observational study that we conducted reported a significant reduction in behavioral disorders of patients during the first 3 months followed by stability. According to the therapists involved in this study, the 3-month format is considered too short to produce perennial benefits; stimulation is often interrupted at the end of the 3 months, which creates a break in management that can be deleterious for patients.

The main objective of this trial is to evaluate the effectiveness of the maintenance of occupational therapy for 4 months beyond the three months provided for in the regulatory framework for the management of demented patients, Measured by the neuropsychiatric inventory (NPI). The secondary objectives will be to study the efficacy on other clinical criteria but also to carry out an economic evaluation of the maintenance of occupational therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with dementia (regardless of etiology) diagnosed or suspected by their physician (general practitioner or specialist) and referred to an Alzheimer specialized team
* Patients with Mini Mental State Examination score> 15
* Patients living at home, in residences for the elderly
* Presence of a non-professional primary caregiver

Exclusion Criteria:

* Patients under 18 years of age;
* Institutionalized or foster care patients;
* Patients who routinely refuse home care;
* Patients with a known severe and unstable general pathology that does not allow patient follow-up;
* Patients already enrolled in another non-drug management trial other than the study;
* Patients whose institutionalization is probable in the short term (within 6 months) or for whom a change of domicile envisaged in the short term and would not allow the carrying out of the follow-up evaluations;
* Patients under tutorship or curatorship, patients unable to express consent;
* Primary caregiver who does not wish to participate in the study or who cannot be available for the follow-up planned for the study;
* Known cognitive deficits or chronic psychosis that do not able patients' follow-up;
* Presence of a primary caregiver with known cognitive or psychiatric disorders (chronic active psychosis) , which doesn't allow the proper conduct of the study;
* Patients who have already benefited from the "occupational" therapy program.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

PRIMARY OUTCOMES:
Neuropsychiatric inventory (NPI) score | NPI score will be measured at 7 months
  Information on the presence, severity and impact of behavioral disorders. NPI is used to evaluate 12 different types of behavior: delusions, apathy, hallucinations, disinhibition, agitation, irritability, depression, aberrant motor behavior, anxiety, night behavior, euphoria, change in appetite and eating behaviors. This inventory is based on the responses obtained by an informed caregiver, preferably living with the patient. The interview is preferably conducted with the caregiver in the patient's absence, to facilitate open discussion of behaviors that may be difficult to describe in the presence of the patient. If a disorder is present, the caregiver should rate the disorder (1: sometimes, 2: quite often, 3: frequently, 4: very frequently) and the severity of the disorder (1: mild, 2: average ; 3: important). An overall score ranging from 0 to 144 is then calculated, a high score representing greater symptoms in presence, frequency and severity.

SECONDARY OUTCOMES:
Neuropsychiatric inventory (NPI) score | at inclusion
  Information on the presence, severity and impact of behavioral disorders. NPI is used to evaluate 12 different types of behavior: delusions, apathy, hallucinations, disinhibition, agitation, irritability, depression, aberrant motor behavior, anxiety, night behavior, euphoria, change in appetite and eating behaviors. This inventory is based on the responses obtained by an informed caregiver, preferably living with the patient. The interview is preferably conducted with the caregiver in the patient's absence, to facilitate open discussion of behaviors that may be difficult to describe in the presence of the patient. If a disorder is present, the caregiver should rate the disorder (1: sometimes, 2: quite often, 3: frequently, 4: very frequently) and the severity of the disorder (1: mild, 2: average ; 3: important). An overall score ranging from 0 to 144 is then calculated, a high score representing greater symptoms in presence, frequency and severity.
Neuropsychiatric inventory (NPI) score | at 3 months
  Information on the presence, severity and impact of behavioral disorders. NPI is used to evaluate 12 different types of behavior: delusions, apathy, hallucinations, disinhibition, agitation, irritability, depression, aberrant motor behavior, anxiety, night behavior, euphoria, change in appetite and eating behaviors. This inventory is based on the responses obtained by an informed caregiver, preferably living with the patient. The interview is preferably conducted with the caregiver in the patient's absence, to facilitate open discussion of behaviors that may be difficult to describe in the presence of the patient. If a disorder is present, the caregiver should rate the disorder (1: sometimes, 2: quite often, 3: frequently, 4: very frequently) and the severity of the disorder (1: mild, 2: average ; 3: important). An overall score ranging from 0 to 144 is then calculated, a high score representing greater symptoms in presence, frequency and severity.
Neuropsychiatric inventory (NPI) score | at 12 months
  Information on the presence, severity and impact of behavioral disorders. NPI is used to evaluate 12 different types of behavior: delusions, apathy, hallucinations, disinhibition, agitation, irritability, depression, aberrant motor behavior, anxiety, night behavior, euphoria, change in appetite and eating behaviors. This inventory is based on the responses obtained by an informed caregiver, preferably living with the patient. The interview is preferably conducted with the caregiver in the patient's absence, to facilitate open discussion of behaviors that may be difficult to describe in the presence of the patient. If a disorder is present, the caregiver should rate the disorder (1: sometimes, 2: quite often, 3: frequently, 4: very frequently) and the severity of the disorder (1: mild, 2: average ; 3: important). An overall score ranging from 0 to 144 is then calculated, a high score representing greater symptoms in presence, frequency and severity.
The functional autonomy measured by the Disability Assessment in Dementia (DAD scale). | at inlcusion
  This scale concerns the activities of the patient in his daily life (dressing, toilet, medication management in particular). It evaluates 5 basic activities and 5 instrumental activities. Each of the 10 activities is broken down into 3 factors entitled: "initiation" ("the patient takes only the initiative of"), "organization" ("he or she plans, organizes the activity"), "effective action" (" the activity is carried out efficiently "). The DAD is completed during an interview with the caregiver. An overall score ranges from 0 to 40, this score is converted to a percentage.
The functional autonomy measured by the Disability Assessment in Dementia (DAD scale). | at 3 months
  This scale concerns the activities of the patient in his daily life (dressing, toilet, medication management in particular). It evaluates 5 basic activities and 5 instrumental activities. Each of the 10 activities is broken down into 3 factors entitled: "initiation" ("the patient takes only the initiative of"), "organization" ("he or she plans, organizes the activity"), "effective action" (" the activity is carried out efficiently "). The DAD is completed during an interview with the caregiver. An overall score ranges from 0 to 40, this score is converted to a percentage.
The functional autonomy measured by the Disability Assessment in Dementia (DAD scale). | at 7 months
  This scale concerns the activities of the patient in his daily life (dressing, toilet, medication management in particular). It evaluates 5 basic activities and 5 instrumental activities. Each of the 10 activities is broken down into 3 factors entitled: "initiation" ("the patient takes only the initiative of"), "organization" ("he or she plans, organizes the activity"), "effective action" (" the activity is carried out efficiently "). The DAD is completed during an interview with the caregiver. An overall score ranges from 0 to 40, this score is converted to a percentage.
The functional autonomy measured by the Disability Assessment in Dementia (DAD scale). | at 12 months
  This scale concerns the activities of the patient in his daily life (dressing, toilet, medication management in particular). It evaluates 5 basic activities and 5 instrumental activities. Each of the 10 activities is broken down into 3 factors entitled: "initiation" ("the patient takes only the initiative of"), "organization" ("he or she plans, organizes the activity"), "effective action" (" the activity is carried out efficiently "). The DAD is completed during an interview with the caregiver. An overall score ranges from 0 to 40, this score is converted to a percentage.
Quality of life measured by the Quality of Life in Alzheimer's Disease scale. | at 3 months
  This 13-item scale explores 6 areas of subjective health: fitness, mood, memory, the patient's relationship with family members, financial hardship, and general health. This tool generates quality of life scores per patient ranging from 13 to 52. This score can be weighted by the answers provided by the caregiver. For this weighting, we multiply the patient score by 2, add the caregiver score and divide by 3 to bring the score back to that of the initial scale.
Quality of life measured by the Quality of Life in Alzheimer's Disease scale. | at 7 months
  This 13-item scale explores 6 areas of subjective health: fitness, mood, memory, the patient's relationship with family members, financial hardship, and general health. This tool generates quality of life scores per patient ranging from 13 to 52. This score can be weighted by the answers provided by the caregiver. For this weighting, we multiply the patient score by 2, add the caregiver score and divide by 3 to bring the score back to that of the initial scale.
Quality of life measured by the Quality of Life in Alzheimer's Disease scale. | at 12 months
  This 13-item scale explores 6 areas of subjective health: fitness, mood, memory, the patient's relationship with family members, financial hardship, and general health. This tool generates quality of life scores per patient ranging from 13 to 52. This score can be weighted by the answers provided by the caregiver. For this weighting, we multiply the patient score by 2, add the caregiver score and divide by 3 to bring the score back to that of the initial scale.
Depression of the patient via the Montgomery-Asberg Depression Rating Scale (MADRS). | at 3 months
  This hetero-evaluation scale is used to assess the depressive symptomatology by exploring 10 components: apparent sadness, expressed sadness, internal tension, sleep reduction, appetite reduction, concentration, lassitude, inability to feel, pessimistic thoughts, suicide ideas. Each component is rated from 0 to 6. The total score ranges from 0 to 60, a high score characterizing a depressive symptomatology.
Depression of the patient via the Montgomery-Asberg Depression Rating Scale (MADRS). | at 7 months
  This hetero-evaluation scale is used to assess the depressive symptomatology by exploring 10 components: apparent sadness, expressed sadness, internal tension, sleep reduction, appetite reduction, concentration, lassitude, inability to feel, pessimistic thoughts, suicide ideas. Each component is rated from 0 to 6. The total score ranges from 0 to 60, a high score characterizing a depressive symptomatology.
Depression of the patient via the Montgomery-Asberg Depression Rating Scale (MADRS). | at 12 months
  This hetero-evaluation scale is used to assess the depressive symptomatology by exploring 10 components: apparent sadness, expressed sadness, internal tension, sleep reduction, appetite reduction, concentration, lassitude, inability to feel, pessimistic thoughts, suicide ideas. Each component is rated from 0 to 6. The total score ranges from 0 to 60, a high score characterizing a depressive symptomatology.
Apathy of the patient via the Apathy inventory. | at 3 months
  This questionnaire that collects information on the presence of apathy in patients suffering from cerebral pathologies. It allows the assessment of three clinical dimensions of apathy: emotional blurring, loss of initiative and loss of interest. The assessment is based on the answers of the accompanying person, and because of this, it can also be carried out in severe deteriorations. The possibility of obtaining the patient's appreciation also makes it possible to evaluate the patient's awareness of his disorders. The evaluation of these 3 dimensions takes into account the frequency (rated from 1 to 4) and the severity of the symptoms (rated from 1 to 3). The score for each dimension is obtained by multiplying these two scores, so that the score for each dimension varies from 0 (absence of the symptom) to 12 (very frequent symptom and of serious gravity)
Apathy of the patient via the Apathy inventory. | at 7 months
  This questionnaire that collects information on the presence of apathy in patients suffering from cerebral pathologies. It allows the assessment of three clinical dimensions of apathy: emotional blurring, loss of initiative and loss of interest. The assessment is based on the answers of the accompanying person, and because of this, it can also be carried out in severe deteriorations. The possibility of obtaining the patient's appreciation also makes it possible to evaluate the patient's awareness of his disorders. The evaluation of these 3 dimensions takes into account the frequency (rated from 1 to 4) and the severity of the symptoms (rated from 1 to 3). The score for each dimension is obtained by multiplying these two scores, so that the score for each dimension varies from 0 (absence of the symptom) to 12 (very frequent symptom and of serious gravity)
Apathy of the patient via the Apathy inventory. | at 12 months
  This questionnaire that collects information on the presence of apathy in patients suffering from cerebral pathologies. It allows the assessment of three clinical dimensions of apathy: emotional blurring, loss of initiative and loss of interest. The assessment is based on the answers of the accompanying person, and because of this, it can also be carried out in severe deteriorations. The possibility of obtaining the patient's appreciation also makes it possible to evaluate the patient's awareness of his disorders. The evaluation of these 3 dimensions takes into account the frequency (rated from 1 to 4) and the severity of the symptoms (rated from 1 to 3). The score for each dimension is obtained by multiplying these two scores, so that the score for each dimension varies from 0 (absence of the symptom) to 12 (very frequent symptom and of serious gravity)
Mortality and institutionalization of patients. | at 3 months
  These events as well as their dates will be collected at each follow-up by psychologists with caregivers, or possibly referring physicians.
Mortality and institutionalization of patients. | at 7 months
  These events as well as their dates will be collected at each follow-up by psychologists with caregivers, or possibly referring physicians.
Mortality and institutionalization of patients. | at 12 months
  These events as well as their dates will be collected at each follow-up by psychologists with caregivers, or possibly referring physicians.
The care processes. | at 3 months
  Treatment (anti-dementia, anti-depressant, antipsychotic), consultation with a medical specialist in the last 3 months, speech therapy, home help and type, perception of Personalized Independence Allowance (APA) and the use of a day care will be collected at each follow-up to determine if maintaining the therapy can influence one or more medical and / or social management processes.
The care processes. | at 7 months
  Treatment (anti-dementia, anti-depressant, antipsychotic), consultation with a medical specialist in the last 3 months, speech therapy, home help and type, perception of Personalized Independence Allowance (APA) and the use of a day care will be collected at each follow-up to determine if maintaining the therapy can influence one or more medical and / or social management processes.
The care processes. | at 12 months
  Treatment (anti-dementia, anti-depressant, antipsychotic), consultation with a medical specialist in the last 3 months, speech therapy, home help and type, perception of Personalized Independence Allowance (APA) and the use of a day care will be collected at each follow-up to determine if maintaining the therapy can influence one or more medical and / or social management processes.
The caregiver burden via the Burden Interview with Zarit | at 3 months
  This questionnaire is composed of 22 items measuring the burden of the caregiver. The score on this questionnaire varies from 0 to 88, a high score characterizing a severe "burden". The questionnaire can also be interpreted qualitatively according to 4 modalities (light, light to moderate, moderate to severe and severe).
The caregiver burden via the Burden Interview with Zarit | at 7 months
  This questionnaire is composed of 22 items measuring the burden of the caregiver. The score on this questionnaire varies from 0 to 88, a high score characterizing a severe "burden". The questionnaire can also be interpreted qualitatively according to 4 modalities (light, light to moderate, moderate to severe and severe).
The caregiver burden via the Burden Interview with Zarit | at 12 months
  This questionnaire is composed of 22 items measuring the burden of the caregiver. The score on this questionnaire varies from 0 to 88, a high score characterizing a severe "burden". The questionnaire can also be interpreted qualitatively according to 4 modalities (light, light to moderate, moderate to severe and severe).
The sense of competence of the caregivers | at 3 months
  This composite questionnaire is constructed based on items from the Zarit scale, and from the Bengtson and Kuypers questionnaire [66]. This 35-item questionnaire covers 3 areas: the consequences of caring involvement in the caregiver's personal life, satisfaction with his or her own performance as a caregiver, and patient satisfaction as a recipient of the caregiver's care.
The sense of competence of the caregivers | at 7 months
  This composite questionnaire is constructed based on items from the Zarit scale, and from the Bengtson and Kuypers questionnaire [66]. This 35-item questionnaire covers 3 areas: the consequences of caring involvement in the caregiver's personal life, satisfaction with his or her own performance as a caregiver, and patient satisfaction as a recipient of the caregiver's care.
The sense of competence of the caregivers | at 12 months
  This composite questionnaire is constructed based on items from the Zarit scale, and from the Bengtson and Kuypers questionnaire [66]. This 35-item questionnaire covers 3 areas: the consequences of caring involvement in the caregiver's personal life, satisfaction with his or her own performance as a caregiver, and patient satisfaction as a recipient of the caregiver's care.
Patient care consumption measured by the RUD Lite scale | at 3 months
  Questionnaire estimating medical and medico-social costs related to patient care. This estimate is based on the assessment of the amount of formal resources (drug treatment, hospitalization, outpatient, day hospital, social services, home care) and informal (care and support provided by the caregiver) implied by the daily care of the patient; the resources are valued economically by using the rates of the health insurance and the hourly costs of the medico-social help at home
Patient care consumption measured by the RUD Lite scale | at 7 months
  Questionnaire estimating medical and medico-social costs related to patient care. This estimate is based on the assessment of the amount of formal resources (drug treatment, hospitalization, outpatient, day hospital, social services, home care) and informal (care and support provided by the caregiver) implied by the daily care of the patient; the resources are valued economically by using the rates of the health insurance and the hourly costs of the medico-social help at home
Patient care consumption measured by the RUD Lite scale | at 12 months
  Questionnaire estimating medical and medico-social costs related to patient care. This estimate is based on the assessment of the amount of formal resources (drug treatment, hospitalization, outpatient, day hospital, social services, home care) and informal (care and support provided by the caregiver) implied by the daily care of the patient; the resources are valued economically by using the rates of the health insurance and the hourly costs of the medico-social help at home
The total cost (health and social) of patient care in each of the groups | at 7 months
  The total cost will be described from the data obtained above for the consumption of care and the management processes
The total cost (health and social) of patient care in each of the groups | at 12 months
  The total cost will be described from the data obtained above for the consumption of care and the management processes
The cost per disorder behavior avoided | at 7 months
The cost per disorder behavior avoided | at 12 months
The cost related to the consequences in terms of quality of life of the patient | at 7 months
The cost related to the consequences in terms of quality of life of the patient | at 12 months

CONTACTS AND LOCATIONS:
Locations (8):
- France (8):
  - Aapam-Ssiad, Blaignan
  - SESAME, Bordeaux
  - Castelsanté, Casteljaloux
  - SSIAD Hauts de garonne, Cenon
  - SSIAD du bassin d'Arcachon, La Teste-de-Buch
  - Vie Santé Merignac, Mérignac
  - AMSADHG, Saint-Savin
  - Equipe Espard, Talence

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pimouguet C, Le Goff M, Wittwer J, Dartigues JF, Helmer C. Benefits of Occupational Therapy in Dementia Patients: Findings from a Real-World Observational Study. J Alzheimers Dis. 2017;56(2):509-517. doi: 10.3233/JAD-160820. PMID 27983551
- [Derived] Pimouguet C, Sitta R, Wittwer J, Hayes N, Petit-Moneger A, Dartigues JF, Helmer C. Maintenance of occupational therapy (OT) for dementia: protocol of a multi-center, randomized controlled and pragmatic trial. BMC Geriatr. 2019 Feb 6;19(1):35. doi: 10.1186/s12877-019-1046-x. PMID 30727947